CLINICAL TRIAL: NCT03265158
Title: Evaluation of Peripheral Blood (PB) Immunophenotyping in the Detection of Bone Marrow Involvement in Cases of Follicular Lymphoma (FL), Mantle Cell Lymphoma (MCL) and Marginal Zone Lymphoma (MZL).
Brief Title: Blood Immunophenotyping in Staging of Indolent B-cell Lymphomas V1.0
Acronym: BMPB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4595
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine whether peripheral blood flow cytometry can reduce or replace invasive bone marrow examinations in patients with slow growing lymphomas.

DETAILED DESCRIPTION:
This study will determine whether peripheral blood flow cytometry can reduce or replace invasive bone marrow examinations in patients with slow growing lymphomas.

Patients with certain types of slow growing (indolent) lymphomas, including the most common sub-type, follicular lymphoma, require a bone marrow examination for staging of their lymphoma. This provides prognostic information and can be important for planning treatment. However, despite the use of local anaesthetic, and in some cases sedation, bone marrow examinations can cause pain and discomfort to patients. Complications are rare but include risk of bleeding, infection and even nerve damage.

Flow cytometry of peripheral blood samples can detect low levels of circulating lymphoma cells. A previous study has demonstrated that detection of lymphoma cells by peripheral blood flow cytometry has a good correlation with bone marrow involvement. This study will seek to find if this correlation is evident in a larger, statistically significant patient cohort. Depending on the study results, invasive and painful bone marrow procedures could potentially be reduced or eliminated in patients with certain slow growing lymphomas. Patients diagnosed with follicular lymphoma, mantle cell lymphoma or marginal zone lymphoma and being treated at the Royal Marsden NHS Foundation Trust will be eligible for this study. Participation in the study will require one peripheral blood sample to be taken before the patient's routine bone marrow biopsy. The study is expected to last between 2 - 3 years for data collection of 108 samples.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18yrs of age
* Able to provide informed written consent
* Patients with a diagnosis of follicular lymphoma, marginal zone lymphoma and mantle cell lymphoma requiring staging or re-staging as part of clinical management
* pre-transplant bone marrow assessment
* High grade transformation associated with the above lymphomas will be allowed.

Exclusion Criteria:

* Patients with a histological diagnosis other than those mentioned above or those diagnosed with 2 or more different lymphomas, excluding transformed lymphoma.
* Patients not fit enough to undergo bone marrow examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with follicular lymphoma (FL), mantle cell lymphoma (MCL) and marginal zone lymphoma (MZL).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of PB flow cytometry compared to BM | 3 years
  The primary outcome measure for this study is the positive predictive value of peripheral blood flow cytometry when compared with bone marrow biopsy in determining bone marrow involvement in patients with FL, MCL and MZL.

SECONDARY OUTCOMES:
Negative predictive value of PB flow cytometry compared to BM | 3 years
  The secondary outcome measures for this study are negative predictive value, sensitivity and specificity of peripheral blood flow cytometry when compared with bone marrow biopsy in determining bone marrow involvement in patients with FL, MCL and MZL.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Iyengar, Principal Investigator — Haematology Consulant, The Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, London, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No